CLINICAL TRIAL: NCT03643120
Title: Gender Dysphoria Among Adolescents
Brief Title: Gender Dysphoria Among Adolescents (Norwegian Title: Kjønnsdysfori Blant Ungdom)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Reidar Schei Jessen, PhD candidate, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/1088/REK sør-øst C
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Intervention Model Description: Qualitative interviews, 15 - 20 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Development of diagnostic typology (Other): One main goal is to Development a typology of sub-types of gender dysphoria.
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Explorative study of gender dysphoria.

SUMMARY:
The aim of this study is to explore how gender dysphoria is experienced among adolescents aged 13 - 18 from a clinical population. The method is qualitative, with a phenomenological approach. Qualitative in-depth data on how gender dysphoria is experienced by the adolescents themselves is lacking in the research literature. As a consequence the within perspective from the clients is lacking. In addition, one aim is to help develop further hypothesis and clinical theory and rationale.

DETAILED DESCRIPTION:
For some children and adolescents their ascribed gender at birth do not match with their gender expression or how they identify later in life. If the mismatch between ascribed gender at birth and gender identity and expression and how the body looks like is associated With distress or discomfort of any kind, this is referred to as gender dysphoria in the Research literature and DSM-V (DSM-V, 2014; Kreukels et al., 2012; Wren, 2014). After initial attempts with so called reparative therapy at changing clients' gender identity in accordance with their ascribed gender at birth, sex reassignment became the treatment of choice to gender dysphoria (Wierckx et al., 2014; Wren, 2014). Since the advent of sophisticated physical treatment like hormonal therapy and surgical techniques, capable of removing certain characteristics of the sexual body, an increasing number of clinics globally have started to offer puberty suppression to pubertal adolescents with gender dysphoria, in order to allow more time before making decisions regarding gender identity. This is referred to as the Dutch model, and the clinical aim is to reduce the pressure the youth are experiencing when the body is developing in a way that creates a lot of distress. Many countries have established special clinics, which focus on development of treatment programs, and there has been a steep increase in number of referrals the last years (Kaltiala-Heino, Sumia, Työläjärvi, & Lindberg, 2015). In Norway, 450 clients were referred to the Norwegian National Unit for Gender Dysphoria and Transsexualism (Nasjonal behandlingstjeneste for transseksualisme, NBTS) in 2016. Half of them were under 18, and the number has been multiplied the last years (Nasjonal behandlingstjeneste for transseksualisme, årsrapport 2016). However, clinical treatment has been initiated without clarifying what gender dysphoria is, how it is experienced by those suffering from it and how it should be understood theoretically. A common concern in the research literature and among clinicians has been that important medical interventions have been utilized while the understanding of gender dysphoria among adolescents and Young adults and its psychological implications could be better understood (Kaltiala-Heino et al., 2015; Wren, 2014). In addition, activists and clients have claimed that their perspectives have been overseen by researchers and clinicians (Wren, 2014). Furthermore, there has been increased attention toward gender dysphoria both nationally and internationally. The aim of this project is to do an interview study in collaboration with chief physician at the NBTS, Ira Haraldsen and a reference group with former clients, in order to produce knowledge on how clients between the ages of 13 and 18 years that are being treated at the NBTS experience the gender dysphoria, how they understand the condition and make sense of their experiences and how it affects their lives. Much of the research on gender dysphoria has been quantitative, based on self report from the clients themselves or reports from health professionals (Drescher & Byne, 2012). This means that the research has focused on predictors of good outcome, and delivered important knowledge on the treatment of gender dysphoria. However, there has not been done much research on the psychological nature of gender dysphoria, what psychosocial consequences this has for the development of gender identity and identity in general and how this is experienced by the young people themselves. There is also a lack of theoretical incorporation of gender dysphoria within the clinical and developmental psychological literature, and a psychological approach to it. Furthermore, studies on the outcome of puberty suppression and sex reassignment have demonstrated that although many adolescents improve mentally after transitioning into an other gender and gender dysphoria ameliorate, many are still suffering from severe psychiatric conditions and psychosocial adjustment (Kaltiala-Heinoet al., 2015). Studies have also demonstrated that adolescents undergoing this treatment is in need of psychological monitoring, but the research on how this should be implemented is lacking (de Vries et al., 2014).

NBTS has been at the forefront internationally implementing the Dutch model. The plan is to interview participants that have been referred to NBTS, consisting of clients that are in different phases of the treatment. The methodological approach will be qualitative and phenomenological, aiming to shed light on how gender dysphoria is experienced subjectively, and focusing on the diversity of presentations rather than searching for general principles. An other important aim is to contribute to theory development, drawing on clinical psychological theories as well as biological and medical knowledge and concepts from gender studies. In relation to this, an aim is to generate hypothesis and stimulate further studies. The collaboration between NBTS and the reference group is an opportunity to fill a gap in the international research between clients and activists one the one hand and researchers and clinicians on the other, and contribute to improved understanding of adolescents suffering from gender dysphoria and how clinicians can help them. This is in line with Standards of Care, the recommendations for treatment of gender dysphoria published by the World Professional Association for Transgender Health. According to this report, the perspectives of people having gender dysphoria are essential to ensure good health care, given the discrimination many are experiencing. Besides, in 2015, the Norwegian Directorate of Health published a report on the health services offered to people with gender dysphoria, named Rett til rett kjønn - helse til alle kjønn, based on the work of an expert group consisting of clinicians, activist and clients. The report concludes that there is a need to do more Research on how gender dysphoria is experienced and what consequences it has for young People living with it. Furthermore, the expert group concludes that there is a need for increased knowledge and awareness of gender dysphoria and how young people living with it should be helped among health professionals working in both specialist and primary health care.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the National Treatment Unit for Transsexuality/Gender dysphoria

Exclusion Criteria:

* Not referred to the National Treatment Unit for Transsexuality/Gender dysphoria

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical sub-types | 2021
  The aim is to develop a typology to describe gender dysphoria.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo university hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
The interviews will we transcribed. Not yet decided whether the transcribed material will be made available.